CLINICAL TRIAL: NCT06159582
Title: eSTEP: An Integrated mHealth Intervention to Engage High-risk Individuals Along the Full PrEP Care Continuum
Acronym: eSTEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Collaborators: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Keith Horvath, Professor, San Diego State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HS-2023-0226
Record Dates: First submitted 2023-11-28; First posted 2023-12-06 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Pre-Exposure Prophylaxis (PrEP)
Keywords: Pre-Exposure Prophylaxis (PrEP); HIV Prevention

STUDY DESIGN:
Intervention Model Description: 2-arm RCT with 2:1 randomization to eSTEP treatment group or usual care control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- eSTEP Treatment Group (Active Comparator): Treatment group participants will be given access to eSTEP (Electronic Support to Engage with PrEP), an mHealth intervention to promote engagement on the full PrEP care continuum tailored to the unique needs of transgender women (TW) and gay, bisexual, and other men who have sex with men (GBMSM), in addition to the usual HIV testing and PrEP clinical care.
  Interventions: Behavioral: eSTEP
- Control Arm (Placebo Comparator): Usual HIV testing and PrEP clinical care
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: eSTEP — eSTEP (Electronic Support to Engage with PrEP) is an mHealth intervention to promote engagement on the full PrEP care continuum and is tailored to the unique needs of GBMSM and TW. eSTEP is a mobile app (eSTEP) intervention with interactive components delivered before in-person HIV testing and PrEP initiation visit and interactive components delivered after PrEP is initiated.
  Arms: eSTEP Treatment Group
Behavioral: Usual Care — Usual HIV testing and PrEP clinical care
  Arms: Control Arm

SUMMARY:
The long-term goal of this research is to develop a theoretically grounded, effective, accessible and sustainable mHealth PrEP care continuum intervention for racially/ethnically diverse transgender women (TW) and gay, bisexual, and other men who have sex with men (GBMSM) disproportionately impacted by the HIV epidemic.

To reach this goal, the investigators will compare study outcomes among persons randomized to use a mobile app (eSTEP) intervention tailored to the unique needs of TW and GBMSM with interactive components delivered before in-person HIV testing and PrEP initiation visit and interactive components delivered after PrEP is initiated. The eSTEP group will be compared to usual HIV testing and PrEP care.

DETAILED DESCRIPTION:
Study Design:

The investigators propose to evaluate the feasibility, acceptability, and preliminary impact of eSTEP in a pilot RCT with transgender women (TW) and gay, bisexual, and other men who have sex with men (GBMSM) who are either PrEP naïve or have not been taking PrEP for at least 3 months, randomized (2:1) to receive either the eSTEP intervention or usual PrEP prevention services, and followed for 6 months with assessments at baseline, 12- and 24-weeks. eSTEP is a mobile application (i.e., app) with interactive PrEP components delivered before in-person HIV testing (at a university-based HIV treatment and prevention clinic) to increase PrEP uptake, and components to optimize PrEP adherence and persistence delivered after the participant tests negative for HIV and agrees to start PrEP. eSTEP will be tailored to the unique needs of TW and GBMSM to optimize its impact and relevance for each group.

eSTEP is grounded in the Information, Motivation, Behavioral Skills model [IMB] and also draws from a model of technology adoption. eSTEP intervention components are:

* HIV Testing and PrEP Information
* Identify and Addressing Barriers to PrEP Uptake and Stigma
* PrEP Eligibility Survey and Preparing to Start PrEP
* HIV Testing Visit Preparation
* Appointment Scheduling
* PrEP Adherence Reminders & Self-monitoring for those who start PrEP
* Adherence Feedback
* PrEP Appointment Reminders
* PrEP and Risk Reduction Information Control arm participants will not be offered the eSTEP mobile app and will receive information about how to schedule their HIV testing appointment at the HIV treatment and prevention clinic on their own (which is the standard procedure for the clinic). Community resources will be also provided electronically to control and treatment arm participants.

Study Sample:

Recruitment will be 120 adult (18 years and older) GBMSM and TW participants (n = 85 GBMSM; n = 35 TW) and will reflect at least 50% Black and/or Latinx participants to ensure that eSTEP is piloted among persons most at risk for HIV. This will allow the investigators to explore differences (e.g. by geder, race and ethnicity) for eSTEP to inform future trials.

Recruitment and Clinical Sites:

Participants will be recruited from a university-based HIV treatment and prevention clinic, as well as in the local San Diego GBMSM and TW communities through the following ways: a) ads on social media sites (e.g., Facebook/Instagram; Grindr) that will link to an online pre-screening survey, b) in-person while attending an HIV testing appointment at the HIV treatment and prevention clinic, c) community recruitment with our existing GBMSM and TW Community Advisory Boards (CABs) and partner community organizations, d) via a part-time recruiter (a peer recruiter or someone with experience in the community).

Enrollment, Randomization and Follow-up Visits:

Study candidates will complete a short online pre-screening survey to assess eligibility on REDCap. Preliminarily eligible participants will complete the enrollment visit over Zoom to verify eligibility and complete online written consent. After informed consent, participants will complete an online 30- to 45-minute baseline survey. All participants will be provided with community resources electronically by the study coordinator and asked to schedule an in-person clinical appointment at the HIV treatment and prevention clinic for routine HIV testing, eligibility and safety lab screening for PrEP as routinely offered in the HIV treatment and prevention clinic. Any participant that receives a positive test for HIV during the trial will receive appropriate post-test counseling and treatment by the HIV treatment and prevention clinic staff. All participants will also be provided 3-4 dried blood spot (DBS) testing kits to self-collect their DBS specimen for the TFV-DP analysis (PrEP adherence) with a detailed instruction sheet and link to a video demonstration of the DBS collect procedure. These kits and the first DBS collection may take place either in person at the HIV treatment and prevention clinic or if necessary, by mail.

Participants will be randomized 2:1 either to the intervention arm (eSTEP and usual care) or to the control arm (HIV testing usual care) using the randomization feature in REDCap. Participants randomized to the treatment arm (eSTEP and usual care) will be guided through setting up their user account and user profile, provided with basic training on how to navigate and use intervention components, and given the opportunity to ask questions. Participants in the treatment arm will have immediate access to eSTEP as part of the initial visit.

Participants will undergo an online 30-45-minute survey at week 12 and week 24. All participants receiving either daily oral or on-demand (2-1-1) PrEP will be asked to complete and submit a DBS specimen at week 12 and week 24 using the kits provided earlier in person at HIV treatment and prevention clinic or by mail and will be seen in-person at the HIV treatment and prevention clinic for usual PrEP care follow-up. Participant survey data will be captured in Qualtrics and, along with clinical study data collected from HIV treatment and prevention clinic HIV testing, and PrEP care appointments, will be captured in our web-based case report forms (CRFs) using REDCap (Research Electronic Data Capture) open software and securely transferred to SDSU via a deidentified file. For treatment arm participants, survey data collection may occur on a mobile device that can access the internet and will be housed on the San Diego State University server.

Study retention protocols involve the use of multiple contact methods including telephone calls, text messages, e-mail reminders, social media, and contact information for a friend/family member - and with permission for the use of each.

Exit Interviews:

10 GBMSM and 10 TW in the eSTEP intervention arm only will be purposively selected (high eSTEP user vs. low user; diversity in race/ethnicity) for a 30-60-minute exit interview to assess their experience in the intervention, suggestions for modifications to the existing interface, suggestions for new features, and changes to any study procedures.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Assigned male sex at birth
* Current male & GBMSM identity OR transfeminine (woman, transgender woman, or non-binary) identification
* Self-reported HIV-negative status
* English-speaking (since the pilot intervention will be developed in English)
* Owner of an Android or iPhone mobile device and access to this phone during the 6-month study.
* Willingness and ability to attend HIV prevention visits at the HIV treatment and prevention clinic.
* Consent to allow study team access to study-relevant PHI
* Eligible for PrEP following CDC guidelines (in the past 6 months had a sexual partner with HIV with unknown or detectable viral load, inconsistently used condoms, and/or was diagnosed with a sexually transmitted infection)
* Has never used PrEP or has not used PrEP in the past 3 months

Exclusion Criteria:

* Was a Community Advisory Board Member or participant in the eSTEP focus groups
* Assigned female or intersex at birth
* Living with HIV
* Already taking PrEP
* Under 18 years old
* Does not own a mobile phone
* Does not speak or read English (since the pilot intervention will be developed in English)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Of 120 participants all assigned male at birth, 85 will identify as men who have sex with men, and 35 will identify as transfeminine (woman, transgender woman, or non-binary)
Enrollment: 116 (Actual)
Dates: Start 2024-04-03 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
PrEP Initiation | Within 24 weeks of enrollment
  Percentage of study participants who initiate PrEP
Protective Levels of PrEP | Throughout the 24 weeks of study participation, starting after PrEP initiation
  Percentage of participants who achieve protective levels of PrEP depending on the type of PrEP participants are taking: 1) if taking daily oral or 2-1-1 PrEP, protective level of PrEP is defined by drug level thresholds in the blood; 2) if taking injectable PrEP, protective level of PrEP is defined by timely (+/- 1 week for the second injection; +/- 2 weeks for any subsequent injection) administration.

SECONDARY OUTCOMES:
PrEP Persistence | Throughout the 24 weeks of study participation, starting after PrEP initiation
  Percentage of participants who achieve PrEP persistence defined as: 1) participant's self-report of currently taking PrEP (daily or 2-1-1) or having received last shot of CAB-LA and 2) has an active prescription for PrEP based on study records.

CONTACTS AND LOCATIONS:
Overall Officials: Keith J Horvath, PhD, Principal Investigator — San Diego State University; Susan J Little, MD, Principal Investigator — University of California, San Diego
Locations (1):
- San Diego State University - Department of Psychology, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No
Will share summary statistics, aggregated data. No deidentified data will be publicly available.

REFERENCES:
- [Background] Wilson IB, Lee Y, Michaud J, Fowler FJ Jr, Rogers WH. Validation of a New Three-Item Self-Report Measure for Medication Adherence. AIDS Behav. 2016 Nov;20(11):2700-2708. doi: 10.1007/s10461-016-1406-x. PMID 27098408
- [Background] Poteat T, Wirtz A, Malik M, Cooney E, Cannon C, Hardy WD, Arrington-Sanders R, Lujan M, Yamanis T. A Gap Between Willingness and Uptake: Findings From Mixed Methods Research on HIV Prevention Among Black and Latina Transgender Women. J Acquir Immune Defic Syndr. 2019 Oct 1;82(2):131-140. doi: 10.1097/QAI.0000000000002112. PMID 31180995
- [Background] Volk JE, Marcus JL, Phengrasamy T, Blechinger D, Nguyen DP, Follansbee S, Hare CB. No New HIV Infections With Increasing Use of HIV Preexposure Prophylaxis in a Clinical Practice Setting. Clin Infect Dis. 2015 Nov 15;61(10):1601-3. doi: 10.1093/cid/civ778. Epub 2015 Sep 1. PMID 26334052
- [Background] Murnane PM, Celum C, Mugo N, Campbell JD, Donnell D, Bukusi E, Mujugira A, Tappero J, Kahle EM, Thomas KK, Baeten JM; Partners PrEP Study Team. Efficacy of preexposure prophylaxis for HIV-1 prevention among high-risk heterosexuals: subgroup analyses from a randomized trial. AIDS. 2013 Aug 24;27(13):2155-60. doi: 10.1097/QAD.0b013e3283629037. PMID 24384592
- [Background] Grant RM, Lama JR, Anderson PL, McMahan V, Liu AY, Vargas L, Goicochea P, Casapia M, Guanira-Carranza JV, Ramirez-Cardich ME, Montoya-Herrera O, Fernandez T, Veloso VG, Buchbinder SP, Chariyalertsak S, Schechter M, Bekker LG, Mayer KH, Kallas EG, Amico KR, Mulligan K, Bushman LR, Hance RJ, Ganoza C, Defechereux P, Postle B, Wang F, McConnell JJ, Zheng JH, Lee J, Rooney JF, Jaffe HS, Martinez AI, Burns DN, Glidden DV; iPrEx Study Team. Preexposure chemoprophylaxis for HIV prevention in men who have sex with men. N Engl J Med. 2010 Dec 30;363(27):2587-99. doi: 10.1056/NEJMoa1011205. Epub 2010 Nov 23. PMID 21091279
- [Background] Camp C, Saberi P. Facilitators and barriers of 2-1-1 HIV pre-exposure prophylaxis. PLoS One. 2021 May 20;16(5):e0251917. doi: 10.1371/journal.pone.0251917. eCollection 2021. PMID 34014998
- [Background] Sewell WC, Powell VE, Mayer KH, Ochoa A, Krakower DS, Marcus JL. Nondaily Use of HIV Preexposure Prophylaxis in a Large Online Survey of Primarily Men Who Have Sex With Men in the United States. J Acquir Immune Defic Syndr. 2020 Jun 1;84(2):182-188. doi: 10.1097/QAI.0000000000002332. PMID 32168169
- [Background] Saberi P, Scott HM. On-Demand Oral Pre-exposure Prophylaxis with Tenofovir/Emtricitabine: What Every Clinician Needs to Know. J Gen Intern Med. 2020 Apr;35(4):1285-1288. doi: 10.1007/s11606-020-05651-2. Epub 2020 Jan 21. PMID 31965523
- [Background] John SA, Whitfield THF, Rendina HJ, Parsons JT, Grov C. Will Gay and Bisexual Men Taking Oral Pre-exposure Prophylaxis (PrEP) Switch to Long-Acting Injectable PrEP Should It Become Available? AIDS Behav. 2018 Apr;22(4):1184-1189. doi: 10.1007/s10461-017-1907-2. PMID 28913659
- [Background] Tolley EE, Zangeneh SZ, Chau G, Eron J, Grinsztejn B, Humphries H, Liu A, Siegel M, Bertha M, Panchia R, Li S, Cottle L, Rinehart A, Margolis D, Jennings A, McCauley M, Landovitz RJ. Acceptability of Long-Acting Injectable Cabotegravir (CAB LA) in HIV-Uninfected Individuals: HPTN 077. AIDS Behav. 2020 Sep;24(9):2520-2531. doi: 10.1007/s10461-020-02808-2. PMID 32052214
- [Background] Whitfield THF, Parsons JT, Rendina HJ. Rates of Pre-exposure Prophylaxis Use and Discontinuation Among a Large U.S. National Sample of Sexual Minority Men and Adolescents. Arch Sex Behav. 2020 Jan;49(1):103-112. doi: 10.1007/s10508-019-01602-z. Epub 2019 Dec 16. PMID 31845148
- [Background] Parsons JT, Rendina HJ, Lassiter JM, Whitfield TH, Starks TJ, Grov C. Uptake of HIV Pre-Exposure Prophylaxis (PrEP) in a National Cohort of Gay and Bisexual Men in the United States. J Acquir Immune Defic Syndr. 2017 Mar 1;74(3):285-292. doi: 10.1097/QAI.0000000000001251. PMID 28187084
- [Background] Wagner GA, Wu KS, Anderson C, Burgi A, Little SJ. Predictors of Human Immunodeficiency Virus Pre-Exposure Prophylaxis (PrEP) Uptake in a Sexual Health Clinic With Rapid PrEP Initiation. Open Forum Infect Dis. 2023 Feb 8;10(3):ofad060. doi: 10.1093/ofid/ofad060. eCollection 2023 Mar. PMID 36968957
- [Background] Matacotta JJ, Rosales-Perez FJ, Carrillo CM. HIV Preexposure Prophylaxis and Treatment as Prevention - Beliefs and Access Barriers in Men Who Have Sex With Men (MSM) and Transgender Women: A Systematic Review. J Patient Cent Res Rev. 2020 Jul 27;7(3):265-274. doi: 10.17294/2330-0698.1737. eCollection 2020 Summer. PMID 32760758
- [Background] Ogunbajo A, Storholm ED, Ober AJ, Bogart LM, Reback CJ, Flynn R, Lyman P, Morris S. Multilevel Barriers to HIV PrEP Uptake and Adherence Among Black and Hispanic/Latinx Transgender Women in Southern California. AIDS Behav. 2021 Jul;25(7):2301-2315. doi: 10.1007/s10461-021-03159-2. Epub 2021 Jan 29. PMID 33515132
- [Background] Koechlin FM, Fonner VA, Dalglish SL, O'Reilly KR, Baggaley R, Grant RM, Rodolph M, Hodges-Mameletzis I, Kennedy CE. Values and Preferences on the Use of Oral Pre-exposure Prophylaxis (PrEP) for HIV Prevention Among Multiple Populations: A Systematic Review of the Literature. AIDS Behav. 2017 May;21(5):1325-1335. doi: 10.1007/s10461-016-1627-z. PMID 27900502
- [Background] Loh KP, Liu J, Ganzhorn S, Sanabria G, Schnall R. Establishing a usability cut-point for the health information technology usability evaluation scale (Health-ITUES). Int J Med Inform. 2022 Apr;160:104713. doi: 10.1016/j.ijmedinf.2022.104713. Epub 2022 Feb 5. PMID 35144102
- [Background] Jacobson TA, Kler JS, Bae Y, Chen J, Ladror DT, Iyer R, Nunes DA, Montgomery ND, Pleil JD, Funk WE. A state-of-the-science review and guide for measuring environmental exposure biomarkers in dried blood spots. J Expo Sci Environ Epidemiol. 2023 Jul;33(4):505-523. doi: 10.1038/s41370-022-00460-7. Epub 2022 Aug 13. PMID 35963945
- [Background] Fisher WA, Fisher JD, Harman J, The information-motivation-behavioral skills model: A general social psychological approach to understanding and promoting health behavior. In Wallston JSKA, ed. Social psychological foundations of health and illness. Blackwell Publishing. 2003; 82-106.